CLINICAL TRIAL: NCT05842031
Title: Assessment of Patient Experience and Needs for Patients Undergoing Invasive Inguinal Lymph Node Procedures for Penile Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0112; NCI-2023-03504 (Registry Identifier: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Penile Cancer
MeSH Terms: conditions — Penile Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Semi-structured interviews: Participants with penile cancer who have undergone invasive inguinal lymph node procedure will be recruited to participate in study via telephone recruitment.
  Interventions: Behavioral: Quality of Life Questionnaires; Behavioral: Patient Educational Needs; Behavioral: Symptom Management

INTERVENTIONS:
Behavioral: Quality of Life Questionnaires — Identify what interventions may be helpful in improving quality of life.
Behavioral: Patient Educational Needs — Identify what interventions may be helpful in improving patient educational needs
Behavioral: Symptom Management — Identify what interventions may be helpful in improving symptom management Improve symptom management

SUMMARY:
To learn more about the patient experience undergoing inguinal (in the groin) lymph node procedures for penile cancer during and after surgery.

DETAILED DESCRIPTION:
Objectives

Primary Objective:

To understand the lived experience of patients undergoing invasive inguinal lymph node procedures.

Secondary Objective:

To determine factors that influence decisions and improve experience for patients who need invasive inguinal lymph node procedures.

ELIGIBILITY:
Inclusion Criteria:

--Patients diagnosed with penile cancer who have undergone invasive inguinal node procedures (ILND and/or DSNB) and are at least 6 months post-procedure

Exclusion Criteria:

* Patient's ≤18 years of age
* Patients who have not undergone invasive surgical procedures involving the inguinal lymph nodes
* Non-English-speaking patients For interviews: people who are physically and/or cognitively incapable of participating in a 60minute telephone interview as determined by a clinical provider or the patient.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: M D Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Decision Regret Scale (DRS) questionnaires | through study completion; an average of 1 year
  Score Scale ranges (1-5)
  1. Strongly Agree
  2. Agree
  3. Agree nor Disagree
  4. Disagree
  5. Strongly Disagree

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Pettaway, BS, MD, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org